CLINICAL TRIAL: NCT05105659
Title: Assessment of Cognitive Functions, Psychological Symptoms, and Quality of Life Among B Thalassemia Patients and Their Clinical Correlates.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alya Mohamed, Resident Physician, Assiut University
Other Study IDs: 45545
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: B Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- B thalassemia Major patients
  Interventions: Diagnostic Test: Wechsler IQ for Adults; Diagnostic Test: MAS (Memory assessment scale); Diagnostic Test: Health-Related Quality of Life (HRQoL); Diagnostic Test: Symptom check list 90; Diagnostic Test: Socioeconomic level
- B thalassemia Intermedia patients
  Interventions: Diagnostic Test: Wechsler IQ for Adults; Diagnostic Test: MAS (Memory assessment scale); Diagnostic Test: Health-Related Quality of Life (HRQoL); Diagnostic Test: Symptom check list 90; Diagnostic Test: Socioeconomic level
- Healthy Controls
  Interventions: Diagnostic Test: Wechsler IQ for Adults; Diagnostic Test: MAS (Memory assessment scale); Diagnostic Test: Health-Related Quality of Life (HRQoL); Diagnostic Test: Symptom check list 90; Diagnostic Test: Socioeconomic level

INTERVENTIONS:
Diagnostic Test: Wechsler IQ for Adults — IQ test that measures the cognitive functions and intelligence using a scale and consists of many subtests assessing verbal and non-verbal performance.
Diagnostic Test: MAS (Memory assessment scale) — tool that uses verbal and the visual tasks to assess memory, recall and cognition. The MAS consists of 12 subtests based on the following 7 memory tasks: Verbal Span, List Learning, Prose memory, Visual Span, Visual Recognition, Visual Reproduction and Names-Faces.
Diagnostic Test: Health-Related Quality of Life (HRQoL) — measures multiple aspects of the individual's life and the impact of the disease and treatment on the individual's life. It does so by assessing the individual's own views and perspective of the care and treatment they are receiving and whether consider it satisfactory or not.
Diagnostic Test: Symptom check list 90 — a well-known scale that is used to identify and assess psychological symptoms. It consists of a 90-item checklist having a 5-point rating scale.
Diagnostic Test: Socioeconomic level — scale for measurement of socioeconomic status in health research in Egypt. The new socioeconomic status scale has 7 domains with a total score of 84. Intra-and inter-observer variability and the internal consistency of the scale were assessed.

SUMMARY:
Multiple studies showed the negative impact thalassemia disease and its therapy have on the cognition of these patients. This study aims to assess and compare the cognition, psychological impact and quality of life among patients with B thalassemia major, requiring regular blood transfusion, patients with B thalassemia intermedia, who don't, and healthy controls. Thus, estimating the role of blood transfusion and hemosiderosis in cognitive impairment, psychological symptoms, and low quality of life in these patients.

DETAILED DESCRIPTION:
Thalassemia is one the most common autosomal recessive haemolytic diseases both worldwide and in the middle east. (1) Beta-thalassemia is a disorder characterized by the congenital absence of the beta chain synthesis of the haemoglobin tetramer, In healthy individuals the haemoglobin chain consists of 2 alpha and 2 beta globin chains, as a result the absence of 2 beta chains in the b thalassemia patients results in clinical symptoms as pallor and failure to thrive. (2,3,4) These patients thus rely on blood transfusions for their entire lives, unless they undergo bone marrow transplant, exposing them to many complications both organically and psychologically. (5) Other patients with b thalassemia whose anaemia doesn't require regular blood transfusion are considered to have B thalassemia intermediate. (6)B thalassemia is among one the most common haemoglobinopathies in Egypt, estimating t 1000/ 1.5 million per year live births born with thalassemia disease. (7) Attention, orientation, memory, gnosis, and executive functions are among some of the cognitive functions that enable an individual to perceive, store, interpret and restore information from the surrounding. (8) Studies have shown that patients with B thalassemia have impairment in most of these cognitive functions in comparison to their healthy counterparts.

psychological problems as stress, anxiety, and depression are some of the psychological disorders that negatively impact the lives of thalassemia patients and may cause multiple comorbidities if not managed properly (9) Quality of life is assessed by focusing on the person's own view of his/her life and his/her well-being taking any conditions or issues that may affect the person's life into consideration. (10) Multiple studies showed the negative impact thalassemia disease and its therapy have on the cognition of these patients. This study aims to assess and compare the cognition, psychological impact and quality of life among patients with B thalassemia major, requiring regular blood transfusion, patients with B thalassemia intermedia, who don't, and healthy controls. Thus, estimating the role of blood transfusion and hemosiderosis in cognitive impairment, psychological symptoms, and low quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Patients diagnosed as B thalassemia major and intermedia by Hb Electrophoresis.

Exclusion Criteria:

* Neurological or any other medical disease.
* IQ less than 70.
* Past history or family history of any psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects: will include three groups: Thalassemia major patients group, Thalassemia intermediate patients group, and healthy control group they will be age and sex matched.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Cognitive functions among B Thalassemia Patients | one year
Assessment of Psychological Symptoms among B Thalassemia Patients | one year
Assessment Quality of life among B Thalassemia Patients | one year